CLINICAL TRIAL: NCT00328289
Title: Effect of Intradialytic Electrical Muscle Stimulation and Passive Leg Mobilisation on Blood Pressure and Dialysis Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S12006
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Hypotension
Keywords: Dialysis associated hypotension; Urea removal
MeSH Terms: conditions — Hypotension

INTERVENTIONS:
Device: transcutaneous muscle stimulation, treadmill

SUMMARY:
Hypothesis: Intradialytic blood pressure and dialysis efficacy (in terms of urea removal) improve under electrical muscle stimulation or passive leg movement on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients able to put legs on a treadmill

Exclusion Criteria:

* Dialysis duration shorter than 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure
Urea removal

SECONDARY OUTCOMES:
Number of hypotensive episodes on dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Uehlinger, Prof, Principal Investigator — Department of Nephrology and Hypertension, University Hospital of Berne
Locations (1):
- Department of Nephrology and Hypertension, University Hospital of Berne, Bern, Canton of Bern, Switzerland